CLINICAL TRIAL: NCT01271192
Title: A Randomized Multicenter Clinical Trial of Direct Surgical Resection Compared to Neoadjuvant Followed by Surgical Resection in Treating Patients With Operable Local Recurrent Carcinoma Of The Rectum
Brief Title: Efficacy and Safety Study of Neoadjuvant in Treating Patients With Resectable Local Recurrent Rectal Cancer
Acronym: NARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Second Military Medical University (Other)
Responsible Party: Ping Lan, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU02
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2010-12

CONDITIONS: Rectal Cancer
Keywords: local recurrent rectal cancer; surgical resection; adjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical resection and adjuvant therapy (Active Comparator): Patients receive surgical resection and undergo FOLFIRI for 12 cycles, from 2-4 weeks after operation. Patients undergo radiotherapy once daily 5 days a week for 5-6 weeks, from 8-12 weeks after operation
  Interventions: Procedure: surgical resection and adjuvant therapy
- Neoadjuvant followed by operation (Experimental): Patients receive neoadjuvant chemoradiotherapy (mFOLFIRI for 5 cycles and undergo radiotherapy as in arm I from the second cycle of FOLFIRI), surgery and FOLFORI for 7 cycles from 2-4 weeks after operation.
  Interventions: Procedure: Neoadjuvant followed by operation

INTERVENTIONS:
Procedure: surgical resection and adjuvant therapy — Postoperative:
  Drug: fluorouracil Given IV continuously, Irinotecan Given IV Radiation: radiation therapy Given 5 days a week for 5-6 weeks
  Arms: Surgical resection and adjuvant therapy
Procedure: Neoadjuvant followed by operation — Preoperative:
  Drug: fluorouracil Given IV continuously,Irinotecan Given IV Radiation: radiation therapy Given 5 days a week for 5-6 weeks
  Postoperative:
  Drug: fluorouracil Given IV continuously,Irinotecan Given IV
  Arms: Neoadjuvant followed by operation

SUMMARY:
RATIONALE: Surgical resection and adjuvant therapy has become the main treatment for resectable local recurrent rectal cancer. However the efficacy and safety of adjuvant therapy is still unknown.

PURPOSE: This randomized multicenter clinical trial is studying surgical resection followed by chemo radiotherapy or neoadjuvant chemo radiotherapy followed by surgery and postoperative chemotherapy, comparing them to see the efficacy and safety, then to investigate the effect of adjuvant chemoradiotherapy for resectable local recurrent rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

- Compare the 5-year survival rate in patients with resectable local recurrent rectal cancer treated with either surgical resection or neoadjuvant.

Secondary

* Compare the side effect of chemo radiotherapy according to the Common Toxicity Criteria(CTC) version 2.0 in patients treated with these regimens.
* Compare the postoperative complications in patients treated with these regimens.
* Compare the recurrent rate in patients treated with these regimens.
* Compare the distant metastatic rate in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter clinical trial. Patients are stratified according to participating center, gender, age. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive surgical resection and undergo FOLFIRI for 12 cycles, from 2-4 weeks after operation. Patients undergo radiotherapy once daily 5 days a week for 5-6 weeks, from 8-12 weeks after operation.
* Arm II: Patients receive neoadjuvant chemoradiotherapy (mFOLFIRI for 5 cycles and undergo radiotherapy as in arm I from the second cycle of FOLFIRI), surgery and FOLFORI for 7 cycles from 2-4 weeks after operation.

After completion of study treatment, patients are followed every 3 months for 2 years, and then every 6 months for at least 3 years.

The side effect of chemo radiotherapy, postoperative complications, recurrent rate, distant metastatic rate and 5-year survival rate will be investigated.

PROJECTED ACCRUAL: A total of 360 patients will be accrued for this study within 5 year.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Adenocarcinoma of the rectum
2. Age:18-80 years old
3. Received curative resection when diagnosed as rectal cancer
4. Local recurrence happened >6 months after operation,without distant metastasis
5. Local recurrent mass is resectable confirmed by surgeon and radiologist 6.15 days prior recruit, meet the following criteria:

   * Hematopoietic
   * Absolute neutrophil count ≥ 1,500/mm^3
   * Platelet count ≥ 100,000/mm^3
   * Hepatic
   * Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
   * Alkaline phosphatase ≤ 2 times ULN
   * AST ≤ 2.5 times ULN
   * ALT ≤ 2.5 times ULN
   * No hepatic disease that would preclude study treatment or follow-up
   * No uncontrolled coagulopathy
   * Renal
   * Creatinine clearance > 50 mL/min
   * No renal disease that would preclude study treatment or follow-up

7.ECOG status: 0～1

Exclusion Criteria:

1. Other rectal cancers (i.e.sarcoma,lymphoma,carcinoid,squamous cell carcinoma,or cloacogenic carcinoma)
2. Synchronous colon cancer
3. Hypersensitivity to fluorouracil
4. No More than 4 weeks since prior participation in any investigational drug study
5. Clear indication of involvement of the pelvic side walls by imaging With distant metastasis
6. History of invasive rectal malignancy, regardless of disease-free interval Fertile patients must use effective contraception
7. Uncontrolled hypertension
8. Cardiovascular disease that would preclude study treatment or follow-up
9. Lack of upper gastrointestinal tract integrity or malabsorption syndrome，active upper gastrointestinal tract bleeding
10. Pregnant or nursing, Fertile patients do not use effective contraception
11. Other malignancy within the past 5 years except effectively treated squamous cell or basal cell skin cancer, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum
12. No psychiatric or addictive disorders, or other conditions that, in the opinion of the investigator, would preclude study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2010-12; Primary Completion 2015-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
5-year disease free survival | 5 years
  Compare the 5-year survival rate in patients with resectable local recurrent rectal cancer treated with either surgical resection or neoadjuvant.

SECONDARY OUTCOMES:
Side effect of chemo radiotherapy, postoperative complications, recurrent rate, distant metastatic rate,biomarkers, quality of life, toxic profile, convenience | 5 years
  * Compare the postoperative complications in patients treated with these regimens
  * Compare the recurrent rate in these patients
  * Compare the distant metastatic rate in these patients
  * Compare preoperative quality of life (QOL) of patients.
  * Compare the toxic effects of these regimens in these patients.
  * Compare the convenience of care in patients treated with these regimens

CONTACTS AND LOCATIONS:
Overall Officials: Ping Lan, M.D., Study Director — Sun Yat-sen University
Locations (1):
- Gastrointestinal Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China